CLINICAL TRIAL: NCT05019183
Title: Clinical Impact and Neuro-functional Substrate of Immersive Virtual Reality Sports Practice on Depression
Acronym: DEPRIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020PBMD05; 2020-A03415-34 (Other: IDRCB)
Record Dates: First submitted 2021-08-19; First posted 2021-08-24 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Physical Conditioning, Human; Tomography, Emission-Computed, Single-Photon

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into 2 arms:
  * Experimental arm: patients will beneficiate from a training program in an immersive environment (virtual reality)
  * Control group: patients will beneficiate from a training program in a real (non-virtual) environment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Patients in the experimental arm will perform 6 indoor rower sessions (30 min each, on Day 1, 2, 3, 8, 9 and 10) during which they will be able to move freely in a virtual environment.
  Interventions: Other: Physical training; Other: Virtual reality; Device: Single-photon emission computed tomography (SPECT); Biological: Metabolomics
- Control arm (Other): Patients in the control arm will perform 6 indoor rower sessions (30 min each, on Day 1, 2, 3, 8, 9 and 10) without being exposed to a virtual environment.
  Interventions: Other: Physical training; Device: Single-photon emission computed tomography (SPECT); Biological: Metabolomics

INTERVENTIONS:
Other: Physical training — The subjects will perform 6 indoor rower sessions (30 min each, on Day 1, 2, 3, 8, 9 and 10) with a target heart rate zone of 60%.
Other: Virtual reality — The subjects will be able to move freely in virtual environments while training on the indoor rower.
  Arms: Experimental arm
Device: Single-photon emission computed tomography (SPECT) — SPECT allows the measurement of cerebral perfusion, reflecting the global synaptic activity, via a 3D acquisition of 20 minutes, 15 minutes after injection of 740 MBq of radiotracers (ECD - Neurolite or HMPAo - Cerestab), with iterative reconstruction. The data will be processed at the voxel scale by the SPM12 software, with analysis of brain connectivity.
Biological: Metabolomics — This qualitative approach will aim to identify pathways that are not known (or have not been explored) to optimize the chances of detecting metabolites present depending on the group (physical activity coupled or not with VR). This method is favorable for biomarker discovery.

SUMMARY:
Depression is a major public health issue due to its frequency (prevalence of 7.5% in adults), its difficulties in therapeutic management (ineffective in 30% of cases and poor compliance) and its societal cost (170 billion euros per year). The most frequent clinical expression is a characterized depressive episode.

Physical activity, through better management of emotions and stress, has been proposed as a complementary therapeutic approach in depression. Studies have shown a decrease in depressive symptoms during a sports program of at least 2 weeks in addition to pharmacological treatment. Similarly, mindfulness meditation, because it reduces ruminations, could also improve the therapeutic management of depression. More recently, virtual reality (VR) exposure therapy has also been proposed in the treatment of anxiety and depression, with a benefit of multisensory stimulation induced by a virtual environment in cognitive and sensory-motor rehabilitation and emotion regulation. However, these therapeutic strategies, in addition to pharmacological treatments, have limits. There is thus a real challenge in designing innovative therapeutic programs for the treatment of depression that encourage motivated practice. A sports activity coupled with immersion in VR could combine the benefits of each of these treatments. With the emergence of new immersive technologies, VR allows the recreation of sensory experiences in an environment close to the ecological context. The use of physical activity on an indoor rower or other sensor-equipped device could thus intensify the psychological benefits of exercise and improve compliance. However, there is a lack of clinical evidence to recommend this coupled therapeutic approach in the additional treatment of depression. This approach is part of the embodied virtual medicine road map.

Furthermore, a better understanding of the biological, metabolomic, and cerebral mechanisms underlying this approach could improve its effectiveness. It would make it possible to propose and evaluate biomarkers for therapeutic and prognostic monitoring of depression. In particular, progress in the field of the "-omics" family includes new tools with great potential. This is more specifically the case of metabolomics. The analysis of metabolites present in the organism or released with natural secretions would allow to constitute a metabolomic signature evolving during the treatment. The interest in characterizing metabolomic biomarkers is an interesting avenue to meet the need to establish a biological diagnosis with quantified values, for better objectivity and follow-up. Functional imaging could also be used to highlight regional activity or connectivity anomalies and markers of response to therapy in relation to biology.

The aim of this work is to determine the clinical impact of physical exercise in VR on a depressive state, and to study in biology, metabolomics and neuroimaging the functional substrates of such a practice in order to understand the mechanisms involved and to propose ways to improve the management of depression.

ELIGIBILITY:
Inclusion Criteria:

* patients between the ages of 18 and 65
* with a diagnosis of characterized depressive episode according to the DSM-5 criteria
* able to practice indoor rower.

Exclusion Criteria:

* Pregnant or breastfeeding women
* With major depression as part of bipolar affective disorder
* Presence of a suicidal risk
* Under Cognitive behavioral therapy or whose medication has been modified in the month preceding enrollment
* History of neurological pathology, head injury or mental retardation
* Presence of an addictive comorbidity
* Presence of a major organic pathology
* Presence of a contraindication to virtual reality exposure
* Presence of a contraindication to SPECT
* Presence of a predisposition to discomfort caused by mobile environments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Change in the Questionnaire Inventory of Depressive Symptomatology (QIDS-SR) depression scale score between Day 1 and Day 10 | From Day 1 to Day 10
  This questionnaire is built on the 9 symptoms used in the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5): sad mood, concentration, self-criticism, suicidal ideation, interest, energy/fatigue, sleep disturbance, decreased/increased appetite or weight, and psychomotor slowing/agitation.
  The total score ranges from 0 to 27 with higher scores meaning higher levels of depression.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge
  - CHU La Conception, Marseille
  - Institut Fresnel, CERIMED, Marseille

IPD SHARING:
Plan to Share IPD: Undecided